CLINICAL TRIAL: NCT01426282
Title: The Effects of Health Education Given by Nurse on Out-patient Compliance in Cardiovascular Diseases Prevention and Treatment in China
Brief Title: The Effects of Health Education in Cardiovascular Diseases Prevention and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lihua Xu (Other)
Responsible Party: Sponsor-Investigator, Lihua Xu, chief nurse in Cardiology, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: JHH 001
Record Dates: First submitted 2011-08-02; First posted 2011-08-31 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Cardiovascular Diseases
Keywords: Out-patient Compliance; Nurse, Heath Education; Cardiovascular Diseases; Treatment and Prevention
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention)
  Interventions: Other: no intervention
- nurse education (Experimental)
  Interventions: Other: health education

INTERVENTIONS:
Other: no intervention — no intervention
  Arms: control
Other: health education — 15 minutes health education given by nurse according to " The Chinese Resident Meals Guide " , "National Revision Committee of the Guidelines of Hypertension Prevention and Control in 2005" , " Guidelines on Prevention and Treatment of Blood Lipid Abnormality in Chinese Adults " , " Guideline for diagnosis and treatment of patients with chronic stable angina "," Guideline for prevention and treatment overweight and obesity in chinese adults "
  Other Names: health education given by nurse
  Arms: nurse education

SUMMARY:
The purpose of this study is to evaluate the effects of health education given by nurse on out-patient compliance in cardiovascular diseases prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

* first diagnosis cardiovascular disease

Exclusion Criteria:

* Severe liver and kidney disease or cancer
* Limb movement disorder
* Cognitive impairment
* History of malignant arrhythmia or severe heart failure patients have a high risk of sudden death
* Diabetes
* Cerebrovascular disease
* History of atherosclerotic disease hospital

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
blood pressure | 1 year
  SBP and DBP
lipid | 1 year
  TC,LDL,TG
Adherence drug administration | 1 year
  Adherence drug administration in one month and in one year
Hospitalization | 1 year
  hospitalization due to cardiovascular and cerebrovascular disease

SECONDARY OUTCOMES:
Exercise time(hours/week) | 1 year
smoking | 1 year
  Number of smoker and Amount of smoke per day
body weight | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- the first college of Harbin Medical University, Harbin, Heilongjiang, China